CLINICAL TRIAL: NCT02182102
Title: A Phase I Open Label Study of Continuous Oral Treatment With BIBF 1120 Together With Pemetrexed in Previously Treated Patients With Non-small Cell Lung Cancer
Brief Title: Dose Escalation of BIBF 1120 Combined With Pemetrexed in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.18
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Pemetrexed

ARMS (1):
- BIBF 1120 + Pemetrexed (Experimental)
  Interventions: Drug: BIBF 1120; Drug: Pemetrexed

INTERVENTIONS:
Drug: BIBF 1120
Drug: Pemetrexed

SUMMARY:
The primary objective was to determine the safety, tolerability and maximum tolerate dose (MTD) of BIBF 1120 in combination with pemetrexed. Secondary objectives were to characterize the pharmacokinetic profiles of BIBF 1120 and pemetrexed and to obtain preliminary anti-tumour efficacy information.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of metastatic, unresectable, or locally advanced NSCLC (non-small cell lung cancer)
* Disease progression during or following one prior platinum-based (including prior neoadjuvant or adjuvant therapy) chemotherapy regimen for advanced disease
* Bi-dimensionally measurable disease by one or more techniques (CT (computed tomography), MRI (magnetic resonance imaging), X-ray)
* Age 18 years or older
* Life expectancy of at least three (3) months
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* Written informed consent that is consistent with ICH-GCP (International Conference on Harmonization - Good Clinical Practice) guidelines

Exclusion Criteria:

* Participation in another clinical study within the past 28 days prior to the start of therapy or concomitantly with this study
* Treatment for NSCLC (except radiotherapy for palliative reasons) within the past 28 days prior to Treatment Day 1 of this trial. All toxicities of the previous therapy must have resolved to baseline prior to Treatment Day 1
* Patient has received more than one prior chemotherapy regimen for advanced disease
* Radiotherapy to an area of measurable disease (unless disease progression had been documented following completion of therapy)
* Patients who are unwilling or unable to take folic acid and vitamin B12 supplementation
* Radiotherapy within 4 weeks prior to Treatment Day 1
* Prior treatment with agents that target the vascular endothelial growth factor (VEGF) pathways, including monoclonal antibody therapy (such as bevacizumab) or tyrosine kinase inhibitors
* Active brain metastases (stable for <28 days, symptomatic, or requiring concurrent steroids or antiepileptic therapy). Patients who have received prior whole brain irradiation and whose brain metastases are stable according to the criteria above will not be excluded
* Centrally located tumors with radiologic evidence (CT or MRI) of local invasion of major blood vessels, with exception of those tumors which have received prior irradiation and are stable
* Cavitary or necrotic tumors
* Sanguinous pleural effusion due to disease or pericardial effusion suspicious for disease
* Other active malignancy diagnosed within the past 3 years (other than non-melanomatous skin cancer)
* Gastrointestinal abnormalities that would interfere with intake or absorption (with exception of patients with gastric esophageal reflux disease controlled with proton pump inhibitors) of the study drug, such as a requirement for intravenous alimentation, prior surgical procedures affecting absorption, treatment for peptic ulcer disease within the last 6 months, active gastrointestinal bleeding unrelated to cancer (as evidenced by either hematemesis, hematochezia, or melena in the past 3 months and without endoscopic documented resolution), or malabsorption syndromes
* Significant cardiovascular disease (i.e., uncontrolled hypertension, myocardial infarction within 6 months, unstable angina, serious cardiac arrhythmia, >2 New York Heart Association (NYHA) Grade 2 congestive heart failure)
* History of hemorrhagic or thrombotic event (including transient ischemic attacks) in the past 12 months or clinically significant hemoptysis in the past 3 months
* Patients receiving any anti-coagulant therapy (including coumadin, heparin, low molecular weight heparin, and aspirin
* Patient has received prior therapy with pemetrexed
* Absolute neutrophil count (ANC) ≤1,500/μl, platelet count ≤100,000/μl, or hemoglobin <9 gm/dL
* Total bilirubin >1.5 mg/dL (26 μmole/L, SI-Unit equivalent), alanine amino transferase (ALT) and/or aspartate amino transferase (AST) ≥1.5 X upper limit of normal (ULN)
* Inadequate renal function determined by a serum creatinine level >1.5 X ULN
* Patient is unable or unwilling to interrupt aspirin or other NSAIDS for a 5-day period (8 days period for long lasting agents like piroxicam)
* Persistent hematuria or proteinuria (more than trace)
* Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast feeding
* Known or suspected active alcohol or drug abuse
* Patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
MTD (maximum tolerated dose) of BIBF 1120 in combination with pemetrexed (500 mg/m2). | up to 126 days
Incidence and intensity of Adverse Events according to the Common Terminology Criteria for Adverse Events (Version 3.0) associated with increasing doses of BIBF 1120. | up to 126 days

SECONDARY OUTCOMES:
AUC0-24 (Area under the plasma concentration-time curve over the dosing interval τ (24 h) following the first dose of uniform intervals τ) | before and up to 6 hours after adminstration in cycle 2
AUC0-tz (AUC over the time interval from zero to the time of the last quantifiable drug concentration) | before and up to 6 hours after adminstration in cycle 2
AUC0-∞ (AUC over the time interval from zero extrapolated to infinity) | before and up to 6 hours after adminstration in cycle 2
%AUCtz-∞ (the percentage of AUC0-∞ that is obtained by extrapolation) | before and 1, 2, 3, 4, 6 hours after first adminstration in cycle 2
Cpre,1 (Pre-dose plasma concentration) | before first administration of BIBF 1120 on day 2 of cycle 2
C24,1 (Plasma concentration at 24 h following the first dose) | 24 hours after the first administration of BIBF 1120 in cycle 2
Cmax (Maximum measured plasma concentration following the first dosing intervals τ) | before and up to 6 hours after adminstration in cycle 2
tmax (Time from dosing to the maximum plasma concentration following the first dosing intervals τ) | before and up to 6 hours after adminstration in cycle 2
λz (Terminal rate constant in plasma) | before and 1, 2, 3, 4, 6 hours after first adminstration in cycle 2
t1/2 (Terminal half-life) | before and 1, 2, 3, 4, 6 hours after first adminstration in cycle 2
MRTpo (Mean residence time after oral administration) | before and 1, 2, 3, 4, 6 hours after first adminstration in cycle 2
CL/F of BIBF 1120 (Apparent clearance) | before and 1, 2, 3, 4, 6 hours after first adminstration of BIBF 1120 in cycle 2
Vz/F of BIBF 1120 (Apparent volume of distribution during the terminal phase) | before and 1, 2, 3, 4, 6 hours after first adminstration of BIBF 1120 in cycle 2
% AUCtz-∞ for pemetrexed | before and 0.25, 1, 2, 4, 6 hours after administration in cycle 2
C24,1 C48,1 (Plasma concentration at 24 h and 48 h following the first dose of treatment cycle | 24 and 28 hours after administration in cycle 2
MRTiv for pemetrexed (Mean residence time after i.v. administration) | before and 0.25, 1, 2, 4, 6 hours after administration in cycle 2
CL (Clearance) for pemetrexed | before and 0.25, 1, 2, 4, 6 hours after administration in cycle 2
Vz for pemetrexed (apparent volume of distribution during the terminal phase following an intravascular dose) | before and 0.25, 1, 2, 4, 6 hours after administration in cycle 2
Vss for pemetrexed (Apparent volume of distribution at steady state) | before and 0.25, 1, 2, 4, 6 hours after administration in cycle 2
Objective tumor response according to the response evaluation criteria in solid tumors (RECIST) | up to 56 months
Duration of objective tumor response (time from best response to onset of tumor progression) | up to 56 months
Time to tumor progression (time from start of treatment to time of documented tumor progression) | up to 56 months